CLINICAL TRIAL: NCT06679829
Title: Phase II Randomized Trial of Population PK Dosed Melphalan With Interleukin-6 Blockade With Siltuximab Vesrus BSA Based Melphalan in Patients With Multiple Myeloma Over Age 60 Undergoing Autologous Stem Cell Transplantation
Brief Title: A Study of Melphalan With or Without Siltuximab in People With Multiple Myeloma Having an Autologous Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-207
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Melphalan; Interleukin-6 Blockade with Siltuximab; Autologous Stem Cell Transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — siltuximab; Melphalan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Siltuximab plus population PK-dosed melphalan (Experimental): For patients randomized to Arm A, the siltuximab, 11 mg/kg, will be administered seven days before and 14 days after autologous hematopoietic stem cell infusion (+/-2 day). Patients will then receive 70mg/m2 of melphalan on Day -2. The melphalan will be infused over 30 minutes. Six peripheral blood samples of 5 ml in lithium heparin tubes will be collected at 5, 15, 30, 40, 75, and 150 minutes after the end of the melphalan infusion for PK testing. The first four time points are +/- 2 min and the last two time points are +/- 5 minutes. The population PK formula in the Insight Rx software will be used to calculate the melphalan dose for Day -1 to achieve a total target area under the curve (AUC) of 13 mg*h/L (+/-1.5). The six PK samples will be collected again after the dose on Day -1 to confirm the total AUC. Patients will receive a minimum of the equivalent of 70mg/m2 and a maximum of the equivalent of 260mg/m2.
  Interventions: Drug: Siltuximab; Drug: Melphalan
- Standard BSA-dosed melphalan (Active Comparator): Patients randomized to Arm B with received Standard of care (SOC) BSA based melphalan dosing at 140 or 200mg/m2 per treating physician on Day -2 and will not receive the siltuximab. The melphalan will be infused over 30 minutes. Six peripheral blood samples of 5 ml in lithium heparin tubes will be collected at 5, 15, 30, 40, 75, and 150 minutes after the end of the melphalan infusion for PK testing. The first four time points are +/- 2 min and the last two time points are +/- 5 minutes.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Siltuximab — 11 mg/kg, will be administered seven days before and 14 days after autologous hematopoietic stem cell infusion (+/-2 day).
  Arms: Siltuximab plus population PK-dosed melphalan
Drug: Melphalan — Arm A: 70mg/m2 of melphalan on Day -2.
  Arm B: SOC BSA based melphalan dosing at 140 or 200mg/m2 per treating physician on Day -2

SUMMARY:
The purpose of this study is to see if siltuximab plus population pharmacokinetic (PK)-dosed melphalan works as well as the usual approach (body surface area [BSA]-dosed melphalan) in people with multiple myeloma (MM) who are receiving an autologous stem cell transplant (ASCT) as part of their standard treatment. The researchers will also see if siltuximab in combination with population PK-dosed melphalan works to decrease symptoms after an ASCT, and will study the safety of siltuximab.

For the run-in, 15 patients will receive siltuximab, 11 mg/kg, seven days before and 14 days after autologous hematopoietic stem cell infusion (+/-2 day).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed symptomatic multiple myeloma undergoing autologous HCT with plan off study for melphalan 140 or 200 mg/m2 undergoing HCT within 12 months of diagnosis.
* At least 60 years of age
* Have at least 3 million x 10^6 CD34+ cells/kg to be infused
* KPS performance status >60% or ECOG Performance Status score of 0-2

Within 6 weeks prior to enrollment:

* Diffusion capacity >45% (adjusted for hemoglobin) as predicted by pulmonary function testing.
* LVEF >45% by MUGA or rest ECHO
* Clinical laboratory values meeting the following criteria

  * Platelet count ≥ 20 x 10^9/L
  * ALT and AST ≤ 2.5 x ULN o Total bilirubin ≤ 2.5 x ULN; except if the elevation is due to Gilbert's syndrome
  * Calculated creatinine clearance > 40 mL/min
* Before enrollment, all women are expected to be not of childbearing potential as they will be age 60+.
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Prior exposure to agents targeting IL-6 or the IL-6 receptor
* Other malignancy within the past 2 years, except for the following if treated and not active: basal cell or nonmetastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or International Federation of Gynecology and Obstetrics (FIGO) Stage 1 carcinoma of the cervix. Prostate cancer under observation may be enrolled after discussion with the MSK Principal Investigator.
* Concurrent medical condition or disease (eg, autoimmune disease, active systemic Infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in the study
* Ischemic heart disease requiring intervention in the prior 3 months or uncontrolled heart failure or an uncontrolled arrhythmiaQTc is >460ms by Fridericia. If they have a right or left bundle branch block or intraventricular conduction delay then exclusion will be for >500ms by Friderica.
* Vaccination with live attenuated vaccines within 4 weeks of first study agent administration
* Clinically significant infection, including known HIV or hepatitis C infection, or known hepatitis B (Hep B) surface antigen positivity. Patients with Hep B Core positivity can be enrolled if the Hep B PCR is negative, and they are on antiviral suppression. Patients with Hepatitis C Ab positive who are PCR negative and have completed Hepatitis C treatment can be enrolled. HIV with negative viral load on HAART can be enrolled.
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 14 days or 5 half lives before enrollment or is currently enrolled in the treatment stage of an investigational study
* Had hospitalization for infection or major surgery (eg, requiring general anesthesia) within 2 weeks before enrollment or have not fully recovered from surgery. Note: subjects with surgical procedures conducted under local anesthesia may participate
* A man who plans to father a child while enrolled in this study or within 3 months after the last dose of study agent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
rate of stringent complete response (sCR) | 100 days
  by modified IMWG based on the day 100 disease evaluation. Urine evaluation will be captured, but response without the urine (unless primary mode of measurement for that patient) will be used for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Gunjan Shah, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm